CLINICAL TRIAL: NCT04742972
Title: PSMA-PET Guided Stereotactic Ablative Body Radiotherapy for Oligometastasis in Metastatic Castration-resistant Prostate Cancer (mCRPC) With Progression on Enzalutamide (PMSABR Study)
Brief Title: Prostate PMSABR Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The lack of well-defined oligometastasis, high disease burden in mCRPC and high sensitivity of PSMA-PET scan, PMSABR study was made with high ambition and the assumption on recruitment was found to be invalid.
Sponsor: Darren Poon (Other)
Responsible Party: Sponsor-Investigator, Darren Poon, Principal Investigator, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PST010
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SABR (Experimental)
  Interventions: Radiation: SABR
- SOC (Placebo Comparator)
  Interventions: Other: SOC

INTERVENTIONS:
Radiation: SABR — SABR is delivered to all sites of oligometastasis with continuation of Enzalutamide. Further oligo-progressive lesions may be treated with SABR if possible. Upon progression at sites not amenable to SABR, the patient may receive any of the options in SOC Arm.
  Arms: SABR
Other: SOC — Three options:
  1. Continuation of Enzalutamide
  2. Observation
  3. Switch to next line treatment
  Arms: SOC

SUMMARY:
In this study, the investigator aim to evaluate the role of PMSA-PET guided SABR on progression free survival (PFS) in patients with oligoprogressive mCRPC with Enzalutamide. The potential improvement in PFS with SABR while continuing the initial-responding Enzalutamide is potentially benefiting to patients in terms of overall disease control.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of prostate adenocarcinoma
* Evidence of stage IV disease (as defined by AJCC criteria) on previous bone, CT, and/or MRI scan
* Ongoing ADT with a gonadotropin-releasing hormone (GnRH) analogue or bilateral orchiectomy (ie, surgical or medical castration) confirmed by testosterone level ≤ 1.73 nmol/L (50 ng/dL) at the screening visit
* ECOG performance score 0-2
* Age ≥ 18
* History/physical examination within 2 weeks prior to registration
* Able to sign informed-consent
* Patient with mCRPC who received Enzalutamide during the past 6-8 weeks and must have been delivered for a total of at least 3 months with an initial ≥50% decline of PSA from baseline.
* Documented disease progression with Enzalutamide as defined by PCWG3 with at least one of the followings:

  1. PSA progression: defined by PSA increase that is ≥ 25% and ≥ 2 ng/mL above the nadir. A minimum of 2 rising PSA levels with an interval of ≥ 1 week between each determination.
  2. Radiographic disease progression in soft tissue based on RECIST 1.1 criteria. Participants whose disease spread is limited to regional pelvic lymph nodes (N1) measuring at least 2 cm in short axis will be considered eligible.
  3. Radiographic disease progression in bone defined as appearance of 2 or more new bone lesions on bone scan
* A maximum of 5 extracranial metastases in any organ system (except brain), with ≤ 4 tumours within any given organ system, confirmed with PSMA PET-CT scan
* All sites of oligometastasis can be safely treated with SABR
* Adequate baseline organ function to allow SABR to all relevant targets
* Participants already receiving agents for the management of skeletal-related events (SREs) are allowed to continue with anti-bone resorptive therapy (including, but not limited to bisphosphonate or receptor activator of nuclear factor kappa ligand inhibitor) if on stable dose for more than 28 days prior to treatment arm assignment

Exclusion Criteria:

* Patients with active cancer other than prostate cancer and non-melanoma skin cancer.
* Prior treatment with docetaxel, another chemotherapy agent or second generation hormonal therapy (e.g. abiraterone acetate or enzalutamide) for metastatic castration-resistant prostate cancer. Prior docetaxel, abiraterone acetate or enzalutamide for metastatic hormone-sensitive prostate cancer is allowed if ≥ 12 months elapsed from last dose of these treatments.
* PSA at inclusion >20 ng/ml
* Serum creatinine and total bilirubin > 3 times the upper limit of normal
* Liver Transaminases > 5-times the upper limit of normal
* Unstable angina and/or congestive heart failure requiring hospitalization, transmural myocardial infarction within the last 6 months, acute bacterial or fungal infection requiring intravenous antibiotics, chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
* Patients with oligometastases that have been previously treated with SABR.
* Serious medical comorbidities precluding radiotherapy, such as ataxia-telangiectasia or scleroderma. For patients with oligoprogressive lesions in the lung or thorax, this includes interstitial lung disease
* Clinical or radiological evidence of spinal cord compression or tumor within 1.5mm of spinal cord on MRI
* Malignant pleural effusion
* Malignant peritoneal disease
* Intra-cranial metastases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
The 6-month progression-Free Survival rate | up to 2 years

SECONDARY OUTCOMES:
Progression-Free Survival | 2 years
Time to progression | 2 years
Overall survival | 2 years
Local control rate of the SABR-treated oligometastasis at 6 months after SABR | up to 2 years
Local control rate of the SABR-treated oligometastasis at 6 months after SABR based on the PERCIST criteria | up to 2 years
QOL (EORTC QLQ-C30) | 2 years
Time to next systemic treatment | 2 years
The number of participants with treatment-related adverse event as assessed by CTCAE v4.0 | 2 years
The proportion of patients in both arms who have AR-V7 (CTCs) | 2 years

IPD SHARING:
Plan to Share IPD: No